CLINICAL TRIAL: NCT03975686
Title: Effects of Neuromuscular Pelvic Realigning Exercises on Pelvic Floor Muscle Function in Continent Subjects: A Randomized Control Trial
Brief Title: Effects of Neuromuscular Pelvic Realigning Exercises on Pelvic Floor Muscle Function in Continent SubjectS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of North Georgia (Other)
Responsible Party: Principal Investigator, Mohammad(Reza) Nourbakhsh, Full Professor, University of North Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNorthGeorgia
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pelvic Floor Muscle Weakness; Stress Urinary Incontinence; Pelvic Asymmetry
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental)
  Interventions: Other: neuromuscual realigning exercise
- control (No Intervention)

INTERVENTIONS:
Other: neuromuscual realigning exercise — neuromuscular realigning exercise
  Arms: intervention

SUMMARY:
The goal of this research study is to investigate the effect of a new neuromuscular approach for correcting pelvic alignment and improving pelvic floor muscle function. Investigators hypothesized that this approach would be significantly superior than no intervention to improve the ability of pelvic floor muscle contraction, measured by transabdominal sonography as bladder base elevation. Participants will be randomized to the intervention and control groups. while intervention group will receive five supervised sessions of pelvic realigning exercises, the control group will receive no intervention. Bladder base elevation will be measured as an indicator of pelvic floor muscle function, before and after one week intervention in both control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

Positive Ober's test

Exclusion Criteria:

* pelvic/low back pain in previous 12 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-08-29 (Estimated)

PRIMARY OUTCOMES:
bladder base elevation | one week
  the ability to contract pelvic floor muscle measured as bladder base elevation by transabdominal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Mahshid A Chehrehrazi, Student, Study Director — University of North Georgia; Mohammad R Nourbakhsh, professor, Principal Investigator — University of North Georgia
Locations (1):
- University of North Georgia, Dahlonega, Georgia, United States

IPD SHARING:
Plan to Share IPD: No